CLINICAL TRIAL: NCT04415697
Title: Identification of Predictive Gene Expression Profile of Sunitinib Rate Response in Metastatic Clear Cell Renal Carcinomas
Brief Title: Identification of Predictive Gene Expression Profile of Sunitinib Response in Metastatic Clear Cell Renal Carcinomas
Status: Completed | Type: Observational
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Andre Octavio Nicolau Sanches, Medical Doctor, Barretos Cancer Hospital
Other Study IDs: BarretosCH-20201
Record Dates: First submitted 2020-05-23; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Kidney Cancer; Biomarkers; Gene Expression
Keywords: Kidney Cancer; Biomarkers; Gene expression; Predictive rate response; Nanostring
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The samples retained in a biobank, with potential for RNA extraction, as genetic material was extracted and stored at - 80 degrees celsius, in the form of a just frozen sample/tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Those who present complete response, partial response, or stable disease, according to RECIST 1.1.
  Interventions: Diagnostic Test: Gene expression test using nanostring technology.
- Not responders: Those who present progression disease according to RECIST 1.1.
  Interventions: Diagnostic Test: Gene expression test using nanostring technology.

INTERVENTIONS:
Diagnostic Test: Gene expression test using nanostring technology. — Evaluation of gene expression profile of a panel with 770 genes related to disease progression using nanostring technology

SUMMARY:
Renal cell carcinoma accounts for 2-3% of all cancers in western countries. Brazilian kidney cancer data show an incidence of 6,270 new cases for 2018. New target-molecular therapies have emerged in recent years for the treatment of metastatic kidney cancer. Due to the heterogeneity of these patients and the lack of specific markers, therapeutic is currently based on clinical and laboratory analysis. The research for predictive biomarkers may better characterize the kidney cancer therapeutic management. The objectives are to identify a predictive gene expression profile in patients with advanced clear cell renal carcinoma treated with first-line sunitinib and correlate it with rate response, seeking to identify a predictive gene expression profile. As secondary objectives, the investigators will compare the gene expression profile found, with global survival and clinical-pathological characteristics. Materials and methods: To determine through systematic data collection the epidemiological profile, clinical-pathological characteristics, response rate, disease free survival and overall survival of 60 patients with metastatic clear cell renal carcinoma who used sunitinib in the first line between 2009 and 2018 at the Barretos Cancer Hospital. For evaluation of gene expression profile, the investigators will use a panel of a panel with 770 genes related to disease progression using nanostring technology.

Keywords: Renal Cell Carcinoma; Sunitinib; Biomarkers; Gene expression; Nanostring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* At least 18 years
* Metastatic clear cell renal carcinoma
* Primary tumors sample of nephrectomy or core biopsy

Exclusion Criteria:

* insufficient sample for molecular analysis
* Patients with no record of treatment response data
* Patients with a history of previous systemic treatment for Metastatic clear cell renal carcinoma
* Patients with second primary synchronic or metachronic tumor undergoing treatment
* Patients having received less than one cycle of sunitinib in the first line
* Patients have received previous adjuvant and/or neoadjuvant treatment with an interval < 1 year between the end of treatment and the diagnosis of metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients at least 18 years with diagnosis of metastatic clear cell renal carcinoma treated with sunitinib in Barretos Cancer Hospital between Jan/2009 and Jan/2018.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Identify differentially expressed genes in two groups of objective response rate. | One year
  Identify differentially expressed genes, through the nanoString platform, in two groups of objective response rate defined using the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Epidemiological characterization of the metastatic clear cell renal carcinoma population treated with sunitinib in the first line, from Barretos Cancer Hospital. | One Year
  Epidemiological characterization of the metastatic clear cell renal carcinoma population treated with sunitinib in the first line, from Barretos Cancer Hospital and correlate with data from differentially expressed genes.

CONTACTS AND LOCATIONS:
Locations (1):
- Andre Octavio Nicolau Sanches, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided